CLINICAL TRIAL: NCT04954937
Title: Convalescent Plasma Donor Vaccine Study: An Observational Antibody Level Study
Brief Title: Convalescent Plasma Donor Vaccine Study An Observational Antibody Level Study.
Acronym: C-VELVET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Blood and Transplant (Other Government)
Responsible Party: Principal Investigator, Lise Jane Estcourt, Haematologist Consultant, NHS Blood and Transplant
Other Study IDs: 21AS0001
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Anti-SARS-CoV-2 antibodies; COVID-19; Convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two EDTA samples will be collected from each donor. First sample will be analysed for SARS-CoV-2 IgG antibodies using EUROimmun assay. A second sample will be analysed for SARS-CoV-2 neutralising antibody testing and ELISA or other immunological assays for anti-S antibodies using SARS-CoV-2 strains.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a need to understand antibody responses following SARS-COV-2 infection and subsequent vaccination.

DETAILED DESCRIPTION:
This is an observational study to determine changes in antibody levels in individuals who have previously donated COVID-19 convalescent plasma (CCP) and have now received at least one dose of a COVID-19 vaccine. At present these donors could no longer donate CCP as their virus-neutralising antibody levels do not reach the level required (Euroimmun of at least 6 IgG signal/control cutoff).

Two blood samples (9 ml total) will be collected at a local NHSBT donor centre to test the levels of the virus-neutralising antibodies in the plasma against different viral strains.

The results of this study will:

1. Determine whether NHSBT will collect CCP or plasma for medicines (PFM) from vaccinated members of the public that could have boosted antibody levels following vaccine administration.
2. Understand if antibody levels rebound to a concentration suitable for CCP and PFM.
3. Provide the evidence to support the use of CCP for the early treatment in COVID (currently under consideration as a collaboration with European partners).
4. Assist in development of recording vaccination status on NHSBT databases of donors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have had a previous SARS-CoV-2 infection
* Individuals who have previously donated COVID-19 convalescent plasma (CCP)
* Received at least one dose of a SARS-CoV-2 vaccine (any type of vaccine)

Exclusion Criteria:

* Not received a SARS-CoV-2 vaccine

Ages: 17 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-10-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Increase in antibody levels post-vaccination assessed via Euroimmun assay | at least 28 days following vaccination
  Euroimmun assay
Increase in antibody levels post-vaccination assessed via Roche IgG assay | at least 28 days following vaccination
  Roche IgG assay
Increase in antibody levels post-vaccination assessed vial live virus neutralization | at least 28 days following vaccination
  Live virus neutralization (SARS-CoV-2 wild type (WT), alpha,beta and delta variants)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Estcourt, MB BChir, DPhil, Principal Investigator — NHS Blood and Transplant
Locations (1):
- NHSBT - Birmingham Donation Centre, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A- Individual participant data will note be shared.